CLINICAL TRIAL: NCT05969782
Title: The Enzen Trial: Comparison of EVAR Outcomes With Endurant Versus Zenith Endoprosthesis: a Prospective Analysis.
Brief Title: The Enzen Trial: Comparison of Evar Endoprosthesis: Endurant Versus Zenith
Acronym: ENZEN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital do Servidor Publico Estadual (Other)
Responsible Party: Principal Investigator, Rafael de Athayde Soares, MD; PhD, Hospital do Servidor Publico Estadual
Other Study IDs: 32380920.5.0000.5463
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Aortic Aneurysm; Aortoiliac Atherosclerosis
Keywords: aneurysm; aortic; aortic disease
MeSH Terms: conditions — Aortic Aneurysm; Aneurysm; Aortic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Endurant II: Patients with aortoiliac aneurysm submitted to EVAR with Endurant II.
  Interventions: Device: EVAR
- Zenith: Patients with aortoiliac aneurysm submitted to EVAR with Zenith.
  Interventions: Device: EVAR

INTERVENTIONS:
Device: EVAR — Endovascular repair of aortoiliac aneurysm using Zenith or Endurant

SUMMARY:
A prospective, non-randomized trial of patients submitted to EVAR for aortoiliac aneursym using Endurant II (Medtronic) or Zenith (Cook).

DETAILED DESCRIPTION:
A prospective, non-randomized trial of patients submitted to EVAR for aortoiliac aneursym using Endurant II (Medtronic) or Zenith (Cook).

The patients will be evaluated in a follow-up, regarding overall mortality rate, perioperative mortality rate and outcomes, such as Endoleaks and reinterventions.

ELIGIBILITY:
Inclusion Criteria: Aortoiliac infra-renal aneurysms.

-

Exclusion Criteria: Thoracoabdominal aortic aneurysms, pararenal and supra-renal aortic aneurysms

* Patients not suitable for EVAR.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAtiens with infra-renal aortoiliac aneurysms submitted to EVAR.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative Mortality rate | 30 days
  Mortality rate

SECONDARY OUTCOMES:
Reinterventions | 2 years
  Reinterventions during follow-up
Endoleaks | 2 years
  Endoleaks during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital do Servidor Público Estadual de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No